CLINICAL TRIAL: NCT04570748
Title: Effect of Capsular Repair on the Outcomes of Direct Anterior Total Hip Arthroplasty.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Murat Sarikas, Recident of orthopaedic surgery, Bezmialem Vakif University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 32495008292
Record Dates: First submitted 2020-07-23; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Coxarthrosis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Direct anterior hip arthroplasty with capsule repair.
  Interventions: Procedure: Capsule repair
- Group B (Active Comparator): Surgery that the surgeon will not perform capsule repair after performing an initial capsulectomy during total hip arthroplasty
  Interventions: Procedure: capsulectomy

INTERVENTIONS:
Procedure: Capsule repair — Direct anterior hip arthroplasty with or without capsule repair
  Arms: Group A
Procedure: capsulectomy — capsulectomy without repair
  Arms: Group B

SUMMARY:
Total hip arthroplasty is a successful surgical procedure performed as a last-line treatment in primary and secondary coxarthrosis.

Recently, the direct anterior approach (DAA) has gained popularity by maintaining abduction force and reducing dislocation rates.

Soft tissue stability in the anterior is increased by adding capsule repair with the preservation of the posterior structures in the DAA.

The degradation of the biological structure of the capsule due to degenerative changes in the end stage coxarthrosis questions the effectiveness of the capsule repair. therefore, the effect of capsule repair on stability is still controversial.

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral or bilateral primary total hip arthroplasty
* Direct anterior surgical approach
* 18 years of age or older
* Avascular necrosis of the hip

Exclusion Criteria:

* Rheumatoid arthritis of the hip
* Revision hip arthroplasty
* Younger than 18 years of age
* Crowe type 3 and 4 coxarthrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Pelvis magnetic resonance ımages(MRI) evaluation of patients who underwent direct anterior total hip arthroplasty | one year
  The new capsule mass will be evaluated by an independent radiologist. adiologist will evaluate the volume of the new capsule structure in cubic millimeter

IPD SHARING:
Plan to Share IPD: No